CLINICAL TRIAL: NCT00254852
Title: A Single Blind, Multi-Center, Randomized, Prospective Clinical Study Comparing Optecure™ Autograft Extender to Autograft Only in Fusion of the Lumbar Spine
Brief Title: Evaluation of Radiographic and Patient Outcomes Following Lumbar Spine Fusion Using Demineralized Bone Matrix (DBM) Mixed With Autograft
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR04-004
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Stenosis; Spondylolisthesis; Degenerative Disc Disease
Keywords: Primary lumbar fusion; Demineralized Bone Matrix; DBM; Optecure; Allograft; Autograft; Lumbar fusion; Interbody fusion; Instrumented fusion; Non-instrumented fusion; Exactech; Spinal fusion
MeSH Terms: conditions — Constriction, Pathologic; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- O (Active Comparator): This treatment arm includes autograft harvested from local bone and / or the iliac crest, supplemented with a demineralized bone matrix (DBM) autograft extender, Optecure.
  Interventions: Procedure: Posterior Lateral Fusion (PLF); Procedure: Anterior Lumbar Interbody Fusion (ALIF); Procedure: Transforaminal lumbar interbody fusion (TLIF); Procedure: Posterior lumbar interbody fusion (PLIF); Procedure: Extreme lateral interbody fusion (XLIF)
- A (Active Comparator): This treatment arm includes autograft harvested from local bone and / or the iliac crest.
  Interventions: Procedure: Posterior Lateral Fusion (PLF); Procedure: Anterior Lumbar Interbody Fusion (ALIF); Procedure: Transforaminal lumbar interbody fusion (TLIF); Procedure: Posterior lumbar interbody fusion (PLIF); Procedure: Extreme lateral interbody fusion (XLIF)

INTERVENTIONS:
Procedure: Posterior Lateral Fusion (PLF) — Posterior lateral fusion (PLF) of the lumbar spine
  Other Names: PLF
Procedure: Anterior Lumbar Interbody Fusion (ALIF) — Anterior lumbar interbody fusion (ALIF)
  Other Names: ALIF
Procedure: Transforaminal lumbar interbody fusion (TLIF) — Transforaminal lumbar interbody fusion (TLIF)
  Other Names: TLIF
Procedure: Posterior lumbar interbody fusion (PLIF) — Posterior lumbar interbody fusion (PLIF)
  Other Names: PLIF
Procedure: Extreme lateral interbody fusion (XLIF) — Extreme lateral interbody fusion (XLIF)
  Other Names: XLIF

SUMMARY:
The purpose of this study is to compare Optecure™ as an autograft extender (treatment) to autograft alone (control) in patients undergoing 1 or 2 level fusion of the lumbar spine(one level is defined as two adjacent vertebrae), L2 and below.

The primary endpoint will be the assessment of fusion by evaluation of x-rays taken following surgery at each visit. The x-ray evaluation will be conducted by a radiologist who is blinded to the type of treatment each patient has received.

Subjects will be seen at 6 weeks, 3 months, 6 months, 12 months, and 24 months postoperative (post-op). Questionnaires and x-rays will be completed at each visit and a computed tomography (CT) scan will be taken at the 12 month visit(and used to aid in assessment of bridging bone, where appropriate).

DETAILED DESCRIPTION:
Autograft (bone taken from one part of the body and placed in another site on the same individual) has long been considered the gold standard for lumbar spine fusion procedures. Unfortunately, there are complications involved with autograft harvest such as donor site morbidity, increased operating time, and limited supply. Therefore, the use of allograft (bone taken from one body and placed into another individual) as a graft extender has become an acceptable practice, especially in fusions of more than one level where larger quantities of graft material are needed.

In this study, comparisons will be made between patients who are randomized to having fusion with an allograft material (Optecure, Exactech, Inc.) mixed with an autograft to those patients who are randomized to having fusion with autograft alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for primary lumbar fusion of 1 or 2 segments, L2 to S1
* Patient is willing to be blindly randomized to treatment or control and remain blinded for 2 years of follow-up
* Patient is at least twenty-one (21) years of age
* Patient is expected to survive at least 2 years beyond surgery
* Patient is willing to participate by complying with pre- and postoperative visit requirements, including: completion of questionnaires, functional performance tests, and radiographs/CT scan
* Patient is willing and able to review and sign a study Informed Consent form

Exclusion Criteria:

* Patient has a mental or physical condition that would invalidate evaluation results
* Patient is pregnant
* Patient is a prisoner
* Patient has a systemic infection or infection at the proposed surgical site
* Patient has osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
* Patient has a disease of bone metabolism
* Patient is undergoing chemotherapy or radiation treatment
* Patient is currently involved in a study of another product for a similar purpose
* Patient requires post-op management with nonsteroidal anti-inflammatory drugs (NSAIDs)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Radiographic evidence of fusion on x-rays taken at each post-op visit | Immediate post-op, 6-week, 3-month, 6-month, 1-year, 2-year

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) completed at each visit | pre-operative, 6-week, 3-month, 6-month, 1-year, 2-year
SF-12 patient health surveys completed at each visit | Pre-operative, 6-week, 3-month, 6-month, 1-year, 2-year
Perceived pain noted on visual analog scales (VAS) at each visit | Pre-operative, 6-week, 3-month, 6-month, 1-year, 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Amir Fayyazi, MD, Principal Investigator — VSAS Orthopedics
Locations (6):
- United States (6):
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - University of California, San Diego, San Diego, California
  - Slocum Dickson Medical Group, New Hartford, New York
  - State University of New York, Upstate Medical University, Syracuse, New York
  - NeuroSpine Solutions, P.C., Bristol, Tennessee
  - Madigan Army Medical Center, Tacoma, Washington